CLINICAL TRIAL: NCT01685749
Title: The Natural History of Human Stingray Injuries
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Robert J Katzer, Emergency Medical Services Fellow, University of California, Irvine
Other Study IDs: HS#2011-8620
Record Dates: First submitted 2012-09-11; First posted 2012-09-14 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Stingray Injury; Marine Envenomation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled participants: The targeted study population will include all people at Seal Beach who have been identified by the Seal Beach Lifeguards to have been stung by a jellyfish over the course of one year who are adults or children whose parent or guardian is present at the time of the injury. Children and pregnant women are included in the group.

SUMMARY:
Stingray injuries can be a hazard shared by many types of beachgoers. Stingrays often lie in the sand and when stepped on by the unsuspecting beachgoer their tail snaps foreword, resulting in a barbed stinger injecting venom into the victim. Little exists in the current literature on the natural history of stingray injuries. Most of the existing literature looks at the incidence of stings, and to a certain extent the demographic of people who seek care. To our knowledge no study has attempted to collect a more inclusive population of those people who are stung and follow them prospectively to determine the incidence of medical intervention, infection, etc.

This study aims to describe and quantify the natural history of stingray injuries and to better understand their time course and medical requirements. The study setting will be Seal Beach, which reports some of the greatest number of annual stingray injuries for any single beach on the pacific coast. Participants will be identified by the Seal Beach lifeguards who are believed to treat the majority of stingray injuries suffered at the beach. Eligible persons will be consented for participation over the phone by research personnel. If enrolled in the study they will receive a phone call by research personnel one week and one month after the injury that will collect information about the symptoms they have experienced and the medical interventions they have received, if any. This study is strictly observational in nature and will not involve any interventions on the part of study personnel or alter the manner in which or types of medical assessments or treatments.

ELIGIBILITY:
Inclusion Criteria:

* People at Seal Beach, California
* People identified by Life guard personnel as being stung by a stingray at Seal Beach
* Adults or
* Children whose parent or guardian are present at the time of the injury

Exclusion Criteria:

* People who have previously been enrolled in the study
* People who the lifeguard believes were stung or bit by a marine organism other than a stingray or a terrestrial organism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The targeted study population will include all people at Seal Beach who have been identified by the Seal Beach Lifeguards to have been stung by a stingray over the course of one year who are adults or children whose parent or guardian is present at the time of the injury. Children and pregnant women are included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence and duration of particular symptoms, medical evaluations, and treatment | up to 30 days from the date of injury
  This study is descriptive in nature. The primary outcome of this study is the understanding of the natural history of stingray injuries and their treatment. This will be achieved using strictly descriptive statistics of the incidence and duration of particular symptoms, medical evaluations, and treatment. Means, proportions, and confidence intervals of these statistics will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
NO IPD will be shared with other researchers